CLINICAL TRIAL: NCT03914950
Title: Evaluation of the Diagnostic Value of TOF-18F-FDG-PET/CT in Patients With Suspected Pancreatic Cancer
Brief Title: TOF-18F-FDG-PET/CT in Patients With Suspected Pancreatic Cancer
Acronym: TOF-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Protokoll TOF-P V1
Record Dates: First submitted 2019-04-02; First posted 2019-04-16 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer; Pancreatitis; IPMN
Keywords: TOF-18F-FDG PET/CT; pancreatic lesions
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis

STUDY DESIGN:
Intervention Model Description: Prospective study with one single group with two kinds of PET/CT imaging (with TOF-reconstruction and without TOF-reconstruction) for each patient.
Masking Description: All parties involved in the clinical trial have knowledge of the interventions assigned to the individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT results with TOF/without TOF (Other): * Diagnostic CT of the abdomen or upper abdomen (in case of already performed diagnostic CT of the abdomen < 2 weeks ago) with 2 phases, 1 - 4 mSv, ca. 20 sec., 1 x
  * Contrast medium (Iodixanol 550 mg/ml) 1 x 1.4 ml/kg body weight i.v. for 40 sec, 1 x if creatinine, GFR, and TSH levels are within the normal range
  * 1 x 500 ml water oral, 1 x
  * Biopsy or FNA (fine-needle aspiration) or operation of the pancreas
  Interventions: Diagnostic Test: PET/CT results with TOF/without TOF

INTERVENTIONS:
Diagnostic Test: PET/CT results with TOF/without TOF — Diagnostic CT of the abdomen or upper abdomen with parenteral contrast medium (Visipaque=Iodixanol) if creatinine, GFR, and TSH levels are within the normal range and oral (water) contrast medium within TOF-18F-FDG PET/CT. In the case of elevated creatine or decreased GFR or TSH levels a diagnostic CT of the abdomen or upper abdomen without contrast medium is performed.
  Biopsy or FNA or operation of the pancreas.

SUMMARY:
Aim of the prospective study is a better differentiation of benign and malignant lesions in the pancreas in patients with suspected pancreatic cancer using images 30 and 90 min p.i. (post injectionen) and a diagnostic CT (computed tomography) scan of the abdomen within the Time of Flight (TOF)-18F-FDG-PET/CT and thus an improvement of the quality of PET/CT findings.

DETAILED DESCRIPTION:
In the course of this the procedure follows the necessary steps of routine treatment:

1. Assignment of the patient with a suspect of pancreatic cancer.
2. Performing time of flight (TOF)-18F-FDG-PET/CT with images 30 min and 90 min p.i.
3. Performing a diagnostic CT of the abdomen with parenteral contrast medium and pancreatic protocol (in case of normal creatinine, GFR, and TSH levels) as well as oral contrast medium (in accordance with the ESUR-guidelines) as part of the PET/CT examination.
4. Routine performance of the operation /fine needle puncture/biopsy
5. Routine histopathological evaluation of the surgical specimen/biopsy

For this study, a diagnostic CT of the abdomen with contrast medium (intravenous as well as oral) and with pancreatic protocol and without parenteral contrast medium in case of elevated creatinine or decreased TSH (thyroid-stimulating hormone) or GFR (glomerular filtration rate) levels is performed additionally within the routinely performed PET/CT for better differentiation of the target organ from adjacent structures. Furthermore, early (30 min p.i.) and delayed (90 min p.i.) images and a TOF-reconstruction following the PET/CT examination (without patient contact) should be performed for better differentiation between inflammatory and malignant lesions of the pancreas. The regional tracer-uptake should now be measured quantitatively by SUV (Standard Uptake Value) in the TOF-PET/CT images over the FDG-accumulating lesions in the pancreas at those two times. In case of an increased FDG-uptake in the early images, the lesion will be assessed as benign/inflammatory and with an increase of the FDG-uptake in the delayed images as malignant. No FDG-uptake in the early as well as in the delayed images will be classified as benign. As a reference standard, the histopathological diagnosis is used. Subsequently, a cut-off value of the SUV should be determined by ROC-analysis.

According to current scientific evidence regarding the characterization of pancreatic masses by means of "Time of Flight"(TOF)-technique, there are no studies in the literature.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected pancreatic cancer

Exclusion Criteria:

* persons under 18 years of age
* patients with blood glucose level ≥160 mg/dl at the time of the PET/CT examination
* patients who will not be operated or biopsied and in which thus there are no histopathological findings of the pancreas
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Stanzel, MD, Principal Investigator — Medical University of Graz, Austria

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will be available apart from the principle investigator only to the statistician who carries out the statistical evaluation of the study.

REFERENCES:
- [Background] Santhosh S, Mittal BR, Bhasin D, Srinivasan R, Rana S, Das A, Nada R, Bhattacharya A, Gupta R, Kapoor R. Role of (18)F-fluorodeoxyglucose positron emission tomography/computed tomography in the characterization of pancreatic masses: experience from tropics. J Gastroenterol Hepatol. 2013 Feb;28(2):255-61. doi: 10.1111/jgh.12068. PMID 23278193
- [Background] Nagamachi S, Nishii R, Wakamatsu H, Mizutani Y, Kiyohara S, Fujita S, Futami S, Sakae T, Furukoji E, Tamura S, Arita H, Chijiiwa K, Kawai K. The usefulness of (18)F-FDG PET/MRI fusion image in diagnosing pancreatic tumor: comparison with (18)F-FDG PET/CT. Ann Nucl Med. 2013 Jul;27(6):554-63. doi: 10.1007/s12149-013-0719-3. Epub 2013 Apr 12. PMID 23580090
- [Result] Stacul F, van der Molen AJ, Reimer P, Webb JA, Thomsen HS, Morcos SK, Almen T, Aspelin P, Bellin MF, Clement O, Heinz-Peer G; Contrast Media Safety Committee of European Society of Urogenital Radiology (ESUR). Contrast induced nephropathy: updated ESUR Contrast Media Safety Committee guidelines. Eur Radiol. 2011 Dec;21(12):2527-41. doi: 10.1007/s00330-011-2225-0. Epub 2011 Aug 25. PMID 21866433

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at one university hospital between February 2014 and January 2019. The first participant was enrolled on February 7, 2014, and the last participant was enrolled in January 2019.
Pre-assignment Details: Of 174 enrolled participants, 120 participants met ALL inclusion criteria having TOF-18F-FDG PET/CT with diagnostic CT of the abdomen or upper abdomen AND biopsy or FNA or operation of the pancreas and were analyzed. Participants not completing the study were excluded and therefore not analyzed (54 participants).
Groups:
- PET/CT Results With TOF/Without TOF: Participants received TOF-18F-FDG PET/CT 30 and 90min p.i. and diagnostic CT of the abdomen or upper abdomen (in case of already performed diagnostic CT of the abdomen < 2 weeks ago) with contrast medium in the case of normal creatinine, GFR, and TSH levels (101 participants). In the case of elevated creatinine or decreased GFR or TSH levels a diagnostic CT without contrast medium was performed (19 participants). After PET/CT examination the participants received a biopsy or FNA (fine-needle aspiration) or operation of the pancreas.
Period: Overall Study
Arm/Group | PET/CT Results With TOF/Without TOF
Started | 174
Completed | 120
Not Completed | 54
Not completed — Physician Decision | 54

BASELINE CHARACTERISTICS:
Population: Participants with biopsy or FNA or operation of the pancreas.
Groups:
- PET/CT Results With TOF/Without TOF: Participants received TOF-18F-FDG PET/CT 30 and 90 min p.i. and diagnostic CT of the abdomen or upper abdomen (in case of already performed diagnostic CT of the abdomen < 2 weeks ago) with contrast medium in case of normal creatinine, GFR, and TSH levels. In the case of elevated creatinine and decreased GFR and TSH levels a diagnostic CT without contrast medium was performed. After PET/CT examination participants received biopsy or FNA or operation of the pancreas.
Arm/Group | PET/CT Results With TOF/Without TOF
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 120
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 120
Type of pancreatic mass [Count of Participants; unit: Participants]
  Solid | 86
  Solid-cystic | 11
  Cystic | 23
History of pancreatitis [Count of Participants; unit: Participants] | 21
Dignity of pancreatic lesions [Count of Participants; unit: Participants]
  Malignant | 85
  Benign | 35
Pathological diagnoses of malignant pancreatic lesions [Count of Participants; unit: Participants] — Population: 85 of 120 participants had malignant pancreatic lesions.
  Participants
    number analyzed (Participants) | 85
    Adenocarcinoma | 70
    Acinuscellcarcinoma | 1
    Diffuse large cell-B-cell lymphoma | 1
    Follicular lymphoma | 1
    Myeloid sarcoma | 1
    Neuroendocrine carcinoma | 1
    Moderately differentiated neuroendocrine tumor (G2 | 2
    IPMN adenocarcinoma invasive | 1
    IPMN carcinoma non-invasive | 2
    Pancreatic intraepithelial neoplasia III(PanINIII) | 4
    Mesenchymal neoplasia | 1
Pathological diagnoses of benign pancreatic lesions [Count of Participants; unit: Participants] — Population: 35 of 120 participants had benign pancreatic lesions.
  Participants
    number analyzed (Participants) | 35
    Acute pancreatitis | 3
    Chronic pancreatitis | 11
    Mucinous cystic neoplasm (MCN) adenoma | 2
    IPMN borderline-lesion | 2
    Serous cyst adenoma | 3
    Benign cyst | 1
    Highly differentiated neuroendocrine tumor | 1
    No indication of malignancy | 12

OUTCOME MEASURES:

1. Primary Outcome: SUVmax (Maximal Standard Uptake Value) Measurement 30 and 90 Min p.i. (Post Injection)
Description: Quantitative measurement of regional tracer uptake by SUVmax in the TOF-PET/CT and standard PET/CT images over the FDG-accumulating lesions in the pancreas 30 and 90min p.i. The histopathological findings (malignant or benign) were assigned to the corresponding SUVmax values of the pancreatic lesions for the calculation of AUC values in ROC analysis. Then AUC values with and without TOF were compared with the DeLong-test to analyze if there is a significant difference in characterization of pancreatic lesions with TOF.
Time Frame: 2 hours
Population: 120 participants meeting ALL inclusion criteria, i.e. completed TOF-18F-FDG PET/CT AND biopsy or FNA or operation were analyzed. 54 participants had TOF-18F-FDG PET/CT but no biopsy or FNA or operation or the tumor was not in the pancreas and were therefore excluded from the study.
Measure: Number; unit: SUVmax
Groups:
- SUVmax TOF 30min p.i.: SUVmax values of the pancreatic lesions with TOF 30min p.i.
- SUVmax Without TOF 30min p.i.: SUVmax values of the pancreatic lesions without TOF 30min p.i.
- SUVmax TOF 90min p.i.: SUVmax values of the pancreatic lesions with TOF 90min p.i.
- SUVmax Without TOF 90min p.i.: SUVmax values of the pancreatic lesions without TOF 90min p.i.
Arm/Group | SUVmax TOF 30min p.i. | SUVmax Without TOF 30min p.i. | SUVmax TOF 90min p.i. | SUVmax Without TOF 90min p.i.
Number analyzed (Participants) | 120 | 120 | 120 | 120
SUVmax | 0.77 | 0.78 | 0.81 | 0.8
Statistical Analysis 1: Comparison: SUVmax TOF 30min p.i. vs SUVmax Without TOF 30min p.i; It was calculated that 118 participants would have at least 90% power to demonstrate an improvement in specificity of 25% (to 70%) with the new method assuming a specificity of the current method of 45% at a prevalence of malignant lesions of 70% (corresponding to 30% benign lesions). Assumptions included a discontinuation rate of 25%; Test type: Other — The calculation of power and sample size is based on a formula that selects the sample size so that the lower limit of the 95% confidence interval by the expected specificity of the new method most probably exceeds the specificity value of the current method. Receiver operating characteristics (ROC) analysis of the values of SUVmax of the early and delayed images with and without TOF of all pancreatic lesions was done in correlation with the histopathological findings; p = 0.78, DeLong-test; The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: SUVmax TOF 90min p.i. vs SUVmax Without TOF 90min p.i; Test type: Other; p = 0.95, DeLong-test; The threshold for statistical significance was p=0.05

2. Primary Outcome: Participants With Increased Tracer Uptake Over the Pancreatic Lesion With and Without TOF
Description: The number of participants with increased tracer uptake over the pancreatic lesion, i.e. the number of pancreatic lesions with increased tracer uptake with and without TOF. One pancreatic lesion per patient was measured.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Increased Tracer Uptake With TOF: The number of participants with increased tracer uptake with TOF in early or delayed or both images.
- Participants With Increased Tracer Uptake Without TOF: The number of participants with increased tracer uptake without TOF in early or delayed or both images.
Arm/Group | Participants With Increased Tracer Uptake With TOF | Participants With Increased Tracer Uptake Without TOF
Number analyzed (Participants) | 120 | 120
Participants | 116 | 101

3. Secondary Outcome: Lesion Size
Description: Lesion or tumor size in cm in the pancreas measured in the diagnostic CT of the abdomen or upper abdomen.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Lesion Size in cm: The lesion size in cm was measured by the radiologist on diagnostic CT.
Arm/Group | Lesion Size in cm
Number analyzed (Participants) | 120
cm | 3.0 (1.67)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- PET/CT Results With TOF/ Without TOF: 101 participants received diagnostic CT of the abdomen/upper abdomen with contrast medium within the PET/CT examination and 19 participants had diagnostic CT of the abdomen or upper abdomen without contrast medium due to elevated creatine or decreased GFR (glomerular filtration rate) or TSH (thyroid-stimulating hormone) levels.
Arm/Group | PET/CT Results With TOF/ Without TOF
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/CT Results With TOF/ Without TOF (N=101)
Hypotensive shock (Cardiac disorders) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0
Convulsion (Nervous system disorders) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET/CT Results With TOF/ Without TOF (N=101)
Severe vomiting (Gastrointestinal disorders) | 0 (0)
Nausea, mild vomiting (Gastrointestinal disorders) | 0 (0)
Marked urticaria (Skin and subcutaneous tissue disorders) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0)
Facial edema (Skin and subcutaneous tissue disorders) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Vasovagal attack (Nervous system disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
The actual discontinuation rate was higher than expected/anticipated. Therefore, the analysis of the primary outcome measure, a difference between AUC values with and without TOF in ROC-analysis, was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03914950/ICF_000.pdf
  • Study Protocol (2013-09-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03914950/Prot_001.pdf
  • Statistical Analysis Plan (2019-03-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT03914950/SAP_002.pdf